CLINICAL TRIAL: NCT03074929
Title: Improving Childhood Obesity-Related Behavior Change Through Better Risk Communication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Davene Wright, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15895
Record Dates: First submitted 2017-03-01; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Obesity, Childhood
Keywords: risk communication
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel risk communication (Experimental): Intervention parents will receive a novel risk communication message via a tablet app. Parents will also receive height, weight, and BMI percentile information typically provided by a provider during well-child visits as usual.
  Interventions: Behavioral: Novel risk communication
- Usual Care (No Intervention): Parents will receive height, weight, and BMI percentile information typically provided by a provider during well-child visits as usual.

INTERVENTIONS:
Behavioral: Novel risk communication — The investigators will develop novel risk communication messages to communicate the risks of childhood obesity to parents of children with obesity. The investigators will consider several novel approaches around message content and framing, but primarily, we propose using microsimulation models to forecast a child's long-term health risks, based on his age, race, gender, BMI, and family history of CVD.
  Arms: Novel risk communication

SUMMARY:
One-third of American children are overweight or obese, leading to an increased risk for cardiovascular disease (CVD), early mortality, and other risks throughout their lifespan relative to normal weight children. In our pilot work, we found that 67-83% of parents underestimate a child's long-term risk of developing cardiovascular disease in adulthood and that parents thought their own child's risks were 13-15% lower than those of a typical child in their community, even controlling for family health and demographic characteristics. Parents were 40 times less likely to predict that their child, rather than a typical child in their community, would be overweight or obese in adulthood. These findings suggest that parents suffer from optimism bias, the tendency to overestimate one's chances of experiencing unlikely positive events. Belief that a child is at increased risk for adverse health outcomes in adulthood could be an important motivator for a family to initiate behavior changes and vice versa.

The overall goal of this research is to develop provider-based risk communication approaches to motivate parents of obese children to engage in behavior change to protect their children from CVD and other obesity-related co-morbidities later in life. Specifically, the investigators will:

1. Develop risk communication methods that providers can use to better convey accurate information about a child's health behaviors, obesity status, and future health risks to parents.
2. Using an online experiment, we will evaluate the impact of new risk communication methods on parental engagement in behavior change.
3. Pilot test the feasibility, acceptability, and impact of new risk communication approaches in pediatric primary care clinics.

This work will give pediatricians novel tools to effectively discuss the long-term consequences of childhood obesity with parents. The findings from this work will inform an interventional trial that will assess the impact of improved risk communication techniques on child behavior change and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* must be a parent of a 5-12 year old child
* child must be a patient at University of Washington Medical Center
* child must have BMI at or above 95th percentile for age and sex
* parent must have home or mobile internet access

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of logging meals in food diary | 7 days
  Frequency of diet monitoring
Quality of food diary | 7 days
  Quality of diet monitoring (i.e. recording 5 or more different foods per day)

SECONDARY OUTCOMES:
Weight class perception (questionnaire) | 7 days
  Does parent perceive child to be Underweight/About the right weight/Overweight/Obese
Anxiety (Perceived Stress Scale) | 7 days
  Perceived Stress Scale
Concern about child health (CAHPS) | 7 days
  In the last 6 months, did you have any questions or concerns about your child's health or health care?

IPD SHARING:
Plan to Share IPD: No